CLINICAL TRIAL: NCT01470612
Title: A MULTI-CENTER, OPEN-LABEL STUDY OF CP-690,550 IN SUBJECTS WITH MODERATE TO SEVERE ULCERATIVE COLITIS
Brief Title: Long-Term Study Of CP-690,550 In Subjects With Ulcerative Colitis
Acronym: OCTAVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3921139; 2011-004581-14 (EudraCT Number); OCTAVEOPEN (Other: Alias Study Number)
Record Dates: First submitted 2011-10-21; First posted 2011-11-11 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; open-label; long term treatment
MeSH Terms: conditions — Colitis, Ulcerative | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CP-690,550 5 mg BID (Experimental): 5 mg BID
  Interventions: Drug: CP-690,550
- CP-690,550 10 mg BID (Experimental): 10 mg BID
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: CP-690,550 — 5 mg tablets, BID, for at least 12 months
  Arms: CP-690,550 5 mg BID
Drug: CP-690,550 — 10 mg tablets, BID, for at least 12 months
  Arms: CP-690,550 10 mg BID

SUMMARY:
This study is an open label, long-term extension study for subjects with moderate to severe ulcerative colitis designed to evaluate long term therapy of CP-690,550.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed induction studies A3921094 or A3921095 and were classified as not meeting clinical response criteria; OR
* Subjects who completed maintenance study A3921096 or who discontinued treatment early in Study A3921096 due to treatment failure.

Exclusion Criteria:

* Subjects who had a major protocol violation in Study A3921094, A3921095 or A3921096.
* Presence of indeterminate colitis, microscopic colitis, ischemic colitis, infectious colitis, or clinical findings suggestive of Crohn's disease.
* Subjects who have had surgery for ulcerative colitis or in the opinion of the investigator, are likely to require surgery for ulcerative colitis during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 944 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2020-08-06 (Actual); Study Completion 2020-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (252):
- United States (75):
  - Alabama Medical Group, P.C., Mobile, Alabama
  - Desert Sun Clinical Research, LLC, Tucson, Arizona
  - Desert Sun Gastroenterology, Tucson, Arizona
  - Desert Sun Surgery Center, Tucson, Arizona
  - Altman Clinical and Translational Research Institute, La Jolla, California
  - Perlman Medical Offices - UC San Diego Health System, La Jolla, California
  - UCSD Medical Center, La Jolla, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Cedars Sinai Surgery Center, Los Angeles, California
  - Alliance Clinical Research, Oceanside, California
  - Center for Endoscopy- Covenant Surgical Partners, Oceanside, California
  - Sharp Rees-Stealy Medical Group, Inc., San Diego, California
  - Clinical Applications Laboratories, Inc, San Diego, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - UCSF Center for Colitis and Crohn's Disease, San Francisco, California
  - Connecticut Clinical Research Institute, Bristol, Connecticut
  - Endoscopy Center of Connecticut, LLC, Guilford, Connecticut
  - Endoscopy Center of Connecticut, LLC, Hamden, Connecticut
  - Gastroenterology Center of Connecticut, PC, Hamden, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Yale New Haven Hospital, New Haven, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - Nature Coast Clinical Research, Inverness, Florida
  - North Florida Gastroenterology Research, LLC, Orange Park, Florida
  - Citrus Ambulatory Surgery Center, Orlando, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Advanced Gastroenterology Center, Port Orange, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Endoscopy Center, Port Orange, Florida
  - Port Orange Urgent Care, Port Orange, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - Atlanta Center for Gastroenterology, P.C., Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Cotton O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Digestive Disease Associates, PA, Catonsville, Maryland
  - Gastrointestinal Diagnostic Center, Catonsville, Maryland
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Howard County GIDC, Columbia, Maryland
  - East Ann Arbor Health and Geriatrics Center -UMHS, Ann Arbor, Michigan
  - Michigan Clinical Research Unit - UMHS, Ann Arbor, Michigan
  - Medical Science Research Building 1 - UMHS, Ann Arbor, Michigan
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Surgical Centers of Michigan, Troy, Michigan
  - Huron Gastroenterology Associates - Center for Digestive Care, Ypsilanti, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - South Jersey Gastroenterology, P.A., Marlton, New Jersey
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - NYU Langone Long Island Clinical Research Associates, Lake Success, New York
  - IBD Center - The Mount Sinai Hospital, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Kornbluth, Legnani, George MD, PC, New York, New York
  - University of Rochester, Rochester, New York
  - Carolina Research, Carolina Digestive Diseases, Greenville, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Baylor College of Medicine- Baylor Medical Center, Houston, Texas
  - McGovern Medical School -The University of Texas Health Science Center at Houston, Houston, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Alpine Medical Group, Salt Lake City, Utah
  - Salt Lake Regional Hospital, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - VCU Health System Digestive Health Center, Richmond, Virginia
  - VCU Health System Endoscopy Suite, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Center for Digestive Health, Milwaukee, Wisconsin
  - Wisconsin Center for Advanced Research - a division of GI Associates, LLC, Milwaukee, Wisconsin
- Australia (7):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Liverpool Hospital eastern Campus, Liverpool, New South Wales
  - Eastern Health, Box Hill Hospital, Box Hill, Victoria
  - Gastroenterology and Hepatology Unit, Clayton, Victoria
- Austria (3):
  - Landeskrankenhaus Innsbruck, Innsbruck
  - Krankenhaus Barmherzige Brueder St. Veit/Glan, Sankt Veit an der Glan
  - AKH Wien, Universitaetsklinik fuer Innere Medizin III, Vienna
- Belgium (4):
  - GZA St Vincentius, Antwerp
  - AZ Groeninge, Kortrijk
  - UZ Leuven (University Hospital Leuven), Campus Gasthuisberg, Leuven
  - H-Hartziekenhuis Roeselare-Menen vzw, Roeselare
- Hospital de Clinicas de Porto Alegre - HCPA, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (9):
  - University of Calgary, Heritage Medical Research Clinic, TRW Building, Calgary, Alberta
  - University of Alberta Hospital - Walter C. Mackenzie Health Sciences Centre, Edmonton, Alberta
  - University of Alberta - Zeidler Ledcor Centre, Edmonton, Alberta
  - McMaster University Medical Center, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Hopital Maisonneuve-Rosemont/Pavillon Rachel-Tourigny, Montreal, Quebec
  - Montreal General Hospital - McGill University Health Care Centre, Montreal, Quebec
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
- Instituto de Coloproctologia ICO S.A.S., Medellín, Antioquia, Colombia
- University Hospital Center Zagreb, Zagreb, Croatia
- Czechia (4):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Klinicke Centrum ISCARE I.V.F., Gastroenterologie, Prague
  - Nemocnice Strakonice, a.s., Interni oddeleni, Strakonice
  - Krajska Zdravotni, A.S.,, Ústí nad Labem
- Denmark (5):
  - Bispebjerg Hospital, Copenhagen, NV
  - Aalborg Hospital, Aalborg
  - Aarhus University Hospital, Aarhus C
  - Hvidovre Hospital, Hvidovre
  - Odense University Hospital, Odense C
- Estonia (2):
  - West Tallinn Central Hospital, Tallinn, Harju
  - Innomedica OU, Tallinn
- France (10):
  - CHU Amiens-Picardie - Hopital Sud, Amiens
  - Hopital Beaujon, Gastroenterologie, MICI et Assistance Nutritive, Clichy
  - CHU de Nantes - Hotel Dieu-Service d'Hepato-Gastroenterologie, Nantes
  - Hôpital Saint Louis - Service d'hepato-gastroenterologie, Paris
  - Hôpital Saint Louis, Paris
  - Hopital Saint Antoine - Service de Gastroenterologie, Paris
  - Hopital Haut-Leveque-CMC Magellan- Unite de Recherche Clinique, Pessac
  - CHU de Reims - Hopital Robert Debre, Reims
  - Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Rangueil, Toulouse
- Germany (8):
  - Universitatsklinikum Schleswig-Holstein, Campus Kiel, Kiel, Schlewig Holstein
  - Universitaetsmedizin Berlin, Charite Campus Virchow-Klinikum, Medizinische Klinik mit, Berlin
  - Universitaesklinikum Halle, Klinik und Poliklinik fuer Innere Medizin I, Halle
  - Medizinische Hochschule Hannover, Hanover
  - Klinikum Lüneburg, Lüneburg
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - University Hospital Munich-Grosshadern, Munich
  - Universitaetsklinikum Ulm, Ulm
- Hungary (12):
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaza; III. Belgyogyaszat - Gasztroenterologia'., Békéscsaba
  - Peterfy Sandor utcai Korhaz-Rendelointezet es Manninger Jeno Orszagos Traumatologiai Intezet, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak I Belgyogyaszati-Gasztroenterologiai Osztaly, Budapest
  - Pannonia Maganorvosi Centrum Kft., Budapest
  - Szent Margit Kórház, III. Belgyógyászati-Gasztroenterológiai Osztály, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza III.sz. Belgyoyaszat Gasztroenterologia, Gyula
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Karolina Korhaz, Mosonmagyaróvár
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, I. Sz. Belgyogyaszati Klinika, Szeged
  - Javorszky Odon Korhaz, Vác
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - The Edith Wolfson Medical Center/Gastroenterology Department, Holon
  - Rabin Medical Center, Beilinson campus, Petah Tikva
- Italy (3):
  - Istituto Clinico Humanitas IRCCS-IBD Center, Rozzano, Milano
  - AOR Villa Sofia-Cervello, Palermo, PA
  - AOU Mater Domini - U.O. Fisiopatologia Digestiva, Catanzaro
- Japan (21):
  - Aichi Medical University Hospital, Nagakute, Aichi-ken
  - National Hospital Organization Hirosaki National Hospital, Hirosaki, Aomori
  - Toho University Sakura Medical Center, Sakura, Chiba
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido P.W.F.A.C Sapporo-Kosei general Hospital, Sapporo, Hokkaido
  - National Hospital Organization Mito Medical Center, Higashi-ibaraki-gun, Ibaraki
  - Sameshima Hospital, Kagoshima, Kagoshima-ken
  - Kuniyoshi Hospital, Kochi, Kochi
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Osaka City University Hospital, Osaka, Osaka
  - Osaka Medical College Hospital, Takatsuki-shi, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Tokyo Medical And Dental University Hospital, Faculty of Medicine, Bunkyo-ku, Tokyo
  - Tokai University Hachioji Hospital, Hachiōji, Tokyo
  - Jikei University Hospital, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Fukuoka University Chikushi Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - The Hospital of Hyogo College of Medicine, Hyōgo
  - Showa University Hospital, Tokyo
- Digestive Diseases Center GASTRO, Riga, Latvia
- Netherlands (4):
  - VU University Medical Center, Amsterdam
  - Academic Medical Center (AMC), Amsterdam
  - University Medical Center Groningen (UMCG), Groningen
  - Leiden University Medical Center, Leiden
- New Zealand (7):
  - Clinical Trials Unit- Tauranga Hospital-Bay of Plenty (BOP) Clinical School, Tauranga, Bay of Plenty
  - Christchurch Hospital, Christchurch, Canterbury
  - North Shore Hospital (Waitemata District Health Board), Auckland
  - Auckland City Hospital, Auckland
  - Southern District Health Board, Dunedin
  - Waikato Hospital, Hamilton
  - P3 Research Limited, Wellington
- Poland (11):
  - Centrum Medyczne Szpital Sw. Rodziny Sp. z o. o., Lodz, Iodzkie
  - Centrum Endoskopii Zabiegowej, Poradnia Chorob Jelitowych, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Gabinet Lekarski - Janusz Rudzinski, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Klinika Chorob Wewnetrznych i Gastroenterologii z Pododdzialem Leczenia Nieswoistych Chorob, Warsaw, Masovian Voivodeship
  - Oddzial Chorob Wewnetrznych i Gastroenterologii, SP ZOZ Wojewodzki Szpital, Bialystok, Podlaskie Voivodeship
  - H-T. Centrum Medyczne - ENDOTERAPIA, Tychy, Silesian Voivodeship
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Oddzial Kliniczny Gastroenterologii Ogolnej i Onkologicznej, Uniwersytecki Szpital Kliniczny nr, Lodz
  - Endoskopia SP. Z O.O., Sopot
  - NZOZ Vivamed, Warsaw
  - Lexmedica, Wroclaw
- Romania (2):
  - Cabinet Particular Policlinic Algomed SRL, Timișoara, Timiș County
  - Spitalul Universitar de Urgenta Bucharest, Medicina Interna II Gastroenterologie, Bucharest
- Russia (10):
  - Federal State Budgetary Institution "State Scientific Centre of Coloproctology n.a. A.N. Ryzhikh", Moscow
  - State budget Healthcare Institution Moscow regional scientific research clinical institute, Moscow
  - State budget Institution of Healthcare Nizhniy Novgorod Regional Clinical Hospital named after N. A., Nizhny Novgorod
  - Municipal Budget Institution of Healthcare of Novosibirsk, Novosibirsk
  - Federal State Budgetary Institution Scientific Research Institute of Physiology and Fundamental, Novosibirsk
  - FSBI "Scientific Research Institute of Physiology and Fundamental Medicine", Novosibirsk
  - Non-State Healthcare Institution "Road Clinical Hospital at the station Samara", Samara
  - Limited Liability Company Medical Company "Hepatolog", Samara
  - Samara Diagnostic center, X-ray Department, Samara
  - State budget institution of healthcare of Yaroslavl region Regional clinical hospital, Yaroslavl
- Serbia (7):
  - Military Medical Academy, Belgrade, Central Serbia
  - Clinical Centre of Serbia Clinic for Gastroenterology and Hepatology, Belgrade
  - Clinical Hospital Center Zvezdara - Clinic for Gastroenterology and Hepatology, Belgrade
  - Clinical Centre of Kragujevac Clinic for Gastroenterology and Hepatology, Kragujevac
  - Clinical Centre of Vojvodina Emergency Internal Medicine Division, Novi Sad
  - Clinical Centre of Vojvodina, Clinic for Gastroenterology and Hepatology, Novi Sad
  - General Hospital Djordje Joanovic, Zrenjanin
- Slovakia (4):
  - Medak s.r.o., Bratislava
  - "KM Management spol. s.r.o.Gastroenterologicke a hepatologicke centrum Nitra, Nitra
  - Poliklinika Libris, Synergy group, a.s.,, Nové Mesto nad Váhom
  - Gastro I., s.r.o., Prešov
- South Africa (5):
  - Chris Hani Baragwanath Academic Hospital, Johannesburg, Gauteng
  - Panorama Medi-Clinic, Cape Town, Western Cape
  - Louis Leipoldt Medical Centre, Cape Town, Western Cape
  - Dr JP Wright, Cape Town, Western Cape
  - Endocare Research Centre, Paarl, Western Cape
- South Korea (7):
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital,, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Corporacio Sanitaria Parc Tauli, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Clinico San Carlos, Madrid
- National Taiwan University Hospital, Taipei, Taiwan
- Ukraine (13):
  - Regional Municipal Institution "Chernivtsi Regional Clinical Hospital", Chernivtsi
  - Regional Municipal Institution 'Chernivtsi Regional Clinical Hospital', Chernivtsi
  - SI 'Institute of Gastroenterology of the NAMS of Ukraine', Dep.-nt of Stomach and Duodenum diseases, Dnipropetrovsk
  - Municipal Healthcare Institution Kharkiv City Clinical Hospital #2, Kharkiv
  - State Institution "L.T. Malaya Therapy Institute of NAMS of Ukraine", Kharkiv
  - Kyiv Municipal Clinical Hospital #18, Proctology Department, Kyiv
  - LTD "St. Paraskeva Medical Center", Lviv
  - Municipal City Clinical Hospital of the Emergency Medical Care, 1-st Therapy Department of hospital,, Lviv
  - Municipal Institution "Odesa Regional Clinical Hospital", polyclinic department, Odesa
  - "Odesa Clinical Hospital for Railway ""Branch of ""Healthcare center of Private JSC ""Ukrainian, Odesa
  - CI of Uzhgorod Regional Rada Uzhgorod Central Regional Hospital". Therapy Department. SHEI Uzhgorod, Uzhhorod
  - Vinnytsia Regional Clinical Hospital for War Veterans, Therapeutics Dept. No. 2, Vinnytsia
  - Minicipal Institution City Hospital #7, Therapeutic Department,, Zaporizhzhia
- United Kingdom (5):
  - Bristol Royal Infirmary, Bristol, England
  - Addenbrooke's Hospital - Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - The North West London Hospitals NHS Trust, Harrow, Middlesex
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk
  - UCLH NIHR Clinical Research Facility, London, W1T 7HA

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Panes J, D'Haens GR, Sands BE, Ng SC, Lawendy N, Kulisek N, Guo X, Wu J, Vranic I, Panaccione R, Vermeire S. Analysis of tofacitinib safety in ulcerative colitis from the completed global clinical developmental program up to 9.2 years of drug exposure. United European Gastroenterol J. 2024 Jul;12(6):793-801. doi: 10.1002/ueg2.12584. Epub 2024 May 22. PMID 38778549
- [Derived] Rubin DT, Torres J, Regueiro M, Reinisch W, Prideaux L, Kotze PG, Tan FH, Gardiner S, Mundayat R, Cadatal MJ, Ng SC. Association Between Smoking Status and the Efficacy and Safety of Tofacitinib in Patients with Ulcerative Colitis. Crohns Colitis 360. 2024 Jan 20;6(1):otae004. doi: 10.1093/crocol/otae004. eCollection 2024 Jan. PMID 38425446
- [Derived] Rubin DT, Salese L, Cohen M, Kotze PG, Woolcott JC, Su C, Mundayat R, Paulissen J, Torres J, Long MD. Presence of risk factors associated with colectomy among patients with ulcerative colitis: a post hoc analysis of data from the tofacitinib OCTAVE ulcerative colitis clinical program. Therap Adv Gastroenterol. 2023 Aug 7;16:17562848231189122. doi: 10.1177/17562848231189122. eCollection 2023. PMID 37560161
- [Derived] Schreiber S, Rubin DT, Ng SC, Peyrin-Biroulet L, Danese S, Modesto I, Guo X, Su C, Kwok KK, Jo H, Chen Y, Yndestad A, Reinisch W, Dubinsky MC. Major Adverse Cardiovascular Events by Baseline Cardiovascular Risk in Patients with Ulcerative Colitis Treated with Tofacitinib: Data from the OCTAVE Clinical Programme. J Crohns Colitis. 2023 Nov 24;17(11):1761-1770. doi: 10.1093/ecco-jcc/jjad104. PMID 37402275
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Lichtenstein GR, Bressler B, Francisconi C, Vermeire S, Lawendy N, Salese L, Sawyerr G, Shi H, Su C, Judd DT, Jones T, Loftus EV. Assessment of Safety and Efficacy of Tofacitinib, Stratified by Age, in Patients from the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2023 Jan 5;29(1):27-41. doi: 10.1093/ibd/izac084. PMID 36342120
- [Derived] Hudesman DP, Torres J, Salese L, Woolcott JC, Mundayat R, Su C, Mosli MH, Allegretti JR. Long-Term Improvement in the Patient-Reported Outcomes of Rectal Bleeding, Stool Frequency, and Health-Related Quality of Life with Tofacitinib in the Ulcerative Colitis OCTAVE Clinical Program. Patient. 2023 Mar;16(2):95-103. doi: 10.1007/s40271-022-00603-w. Epub 2022 Nov 7. PMID 36336750
- [Derived] Biedermann L, Dubinsky MC, Vermeire S, Fellmann M, Gardiner S, Hur P, Mundayat R, Panes J, Rubin DT. Health-Related Quality of Life Outcomes With Tofacitinib Treatment in Patients With Ulcerative Colitis in the Open-Label Extension Study, OCTAVE Open. Inflamm Bowel Dis. 2023 Sep 1;29(9):1370-1379. doi: 10.1093/ibd/izac222. PMID 36242764
- [Derived] Sandborn WJ, D'Haens GR, Sands BE, Panaccione R, Ng SC, Lawendy N, Kulisek N, Modesto I, Guo X, Mundayat R, Su C, Vranic I, Panes J. Tofacitinib for the Treatment of Ulcerative Colitis: An Integrated Summary of up to 7.8 Years of Safety Data from the Global Clinical Programme. J Crohns Colitis. 2023 Apr 3;17(3):338-351. doi: 10.1093/ecco-jcc/jjac141. PMID 36124702
- [Derived] Loftus EV, Baumgart DC, Gecse K, Kinnucan JA, Connelly SB, Salese L, Su C, Kwok KK, Woolcott JC, Armuzzi A. Clostridium difficile Infection in Patients with Ulcerative Colitis Treated with Tofacitinib in the Ulcerative Colitis Program. Inflamm Bowel Dis. 2023 May 2;29(5):744-751. doi: 10.1093/ibd/izac139. PMID 35792493
- [Derived] Winthrop KL, Vermeire S, Long MD, Panes J, Ng SC, Kulisek N, Mundayat R, Lawendy N, Vranic I, Modesto I, Su C, Melmed GY. Long-term Risk of Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2023 Jan 5;29(1):85-96. doi: 10.1093/ibd/izac063. PMID 35648151
- [Derived] Dubinsky MC, Magro F, Steinwurz F, Hudesman DP, Kinnucan JA, Ungaro RC, Neurath MF, Kulisek N, Paulissen J, Su C, Ponce de Leon D, Regueiro M. Association of C-reactive Protein and Partial Mayo Score With Response to Tofacitinib Induction Therapy: Results From the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2023 Jan 5;29(1):51-61. doi: 10.1093/ibd/izac061. PMID 35380664
- [Derived] Feagan BG, Khanna R, Sandborn WJ, Vermeire S, Reinisch W, Su C, Salese L, Fan H, Paulissen J, Woodworth DA, Niezychowski W, Sands BE. Agreement between local and central reading of endoscopic disease activity in ulcerative colitis: results from the tofacitinib OCTAVE trials. Aliment Pharmacol Ther. 2021 Dec;54(11-12):1442-1453. doi: 10.1111/apt.16626. Epub 2021 Oct 6. PMID 34614208
- [Derived] Panes J, Vermeire S, Dubinsky MC, Loftus EV, Lawendy N, Wang W, Salese L, Su C, Modesto I, Guo X, Colombel JF. Efficacy and Safety of Tofacitinib Re-treatment for Ulcerative Colitis After Treatment Interruption: Results from the OCTAVE Clinical Trials. J Crohns Colitis. 2021 Nov 8;15(11):1852-1863. doi: 10.1093/ecco-jcc/jjab065. PMID 33884415
- [Derived] Sandborn WJ, Peyrin-Biroulet L, Sharara AI, Su C, Modesto I, Mundayat R, Gunay LM, Salese L, Sands BE. Efficacy and Safety of Tofacitinib in Ulcerative Colitis Based on Prior Tumor Necrosis Factor Inhibitor Failure Status. Clin Gastroenterol Hepatol. 2022 Mar;20(3):591-601.e8. doi: 10.1016/j.cgh.2021.02.043. Epub 2021 Mar 6. PMID 33684552
- [Derived] Curtis JR, Regueiro M, Yun H, Su C, DiBonaventura M, Lawendy N, Nduaka CI, Koram N, Cappelleri JC, Chan G, Modesto I, Lichtenstein GR. Tofacitinib Treatment Safety in Moderate to Severe Ulcerative Colitis: Comparison of Observational Population Cohort Data From the IBM MarketScan(R) Administrative Claims Database With Tofacitinib Trial Data. Inflamm Bowel Dis. 2021 Aug 19;27(9):1394-1408. doi: 10.1093/ibd/izaa289. PMID 33324993
- [Derived] Sandborn WJ, Peyrin-Biroulet L, Quirk D, Wang W, Nduaka CI, Mukherjee A, Su C, Sands BE. Efficacy and Safety of Extended Induction With Tofacitinib for the Treatment of Ulcerative Colitis. Clin Gastroenterol Hepatol. 2022 Aug;20(8):1821-1830.e3. doi: 10.1016/j.cgh.2020.10.038. Epub 2020 Oct 27. PMID 33127596
- [Derived] Colombel JF, Osterman MT, Thorpe AJ, Salese L, Nduaka CI, Zhang H, Lawendy N, Friedman GS, Quirk D, Su C, Reinisch W. Maintenance of Remission With Tofacitinib Therapy in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2022 Jan;20(1):116-125.e5. doi: 10.1016/j.cgh.2020.10.004. Epub 2020 Oct 9. PMID 33039585
- [Derived] Sands BE, Colombel JF, Ha C, Farnier M, Armuzzi A, Quirk D, Friedman GS, Kwok K, Salese L, Su C, Taub PR. Lipid Profiles in Patients With Ulcerative Colitis Receiving Tofacitinib-Implications for Cardiovascular Risk and Patient Management. Inflamm Bowel Dis. 2021 May 17;27(6):797-808. doi: 10.1093/ibd/izaa227. PMID 32870265
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Lichtenstein GR, Rogler G, Ciorba MA, Su C, Chan G, Pedersen RD, Lawendy N, Quirk D, Nduaka CI, Thorpe AJ, Panes J. Tofacitinib, an Oral Janus Kinase Inhibitor: Analysis of Malignancy (Excluding Nonmelanoma Skin Cancer) Events Across the Ulcerative Colitis Clinical Program. Inflamm Bowel Dis. 2021 May 17;27(6):816-825. doi: 10.1093/ibd/izaa199. PMID 32766762
- [Derived] Sands BE, Armuzzi A, Marshall JK, Lindsay JO, Sandborn WJ, Danese S, Panes J, Bressler B, Colombel JF, Lawendy N, Maller E, Zhang H, Chan G, Salese L, Tsilkos K, Marren A, Su C. Efficacy and safety of tofacitinib dose de-escalation and dose escalation for patients with ulcerative colitis: results from OCTAVE Open. Aliment Pharmacol Ther. 2020 Jan;51(2):271-280. doi: 10.1111/apt.15555. Epub 2019 Oct 29. PMID 31660640
- [Derived] Sandborn WJ, Panes J, Sands BE, Reinisch W, Su C, Lawendy N, Koram N, Fan H, Jones TV, Modesto I, Quirk D, Danese S. Venous thromboembolic events in the tofacitinib ulcerative colitis clinical development programme. Aliment Pharmacol Ther. 2019 Nov;50(10):1068-1076. doi: 10.1111/apt.15514. Epub 2019 Oct 9. PMID 31599001
- [Derived] Sands BE, Taub PR, Armuzzi A, Friedman GS, Moscariello M, Lawendy N, Pedersen RD, Chan G, Nduaka CI, Quirk D, Salese L, Su C, Feagan BG. Tofacitinib Treatment Is Associated With Modest and Reversible Increases in Serum Lipids in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2020 Jan;18(1):123-132.e3. doi: 10.1016/j.cgh.2019.04.059. Epub 2019 May 8. PMID 31077827
- [Derived] Sandborn WJ, Panes J, D'Haens GR, Sands BE, Su C, Moscariello M, Jones T, Pedersen R, Friedman GS, Lawendy N, Chan G. Safety of Tofacitinib for Treatment of Ulcerative Colitis, Based on 4.4 Years of Data From Global Clinical Trials. Clin Gastroenterol Hepatol. 2019 Jul;17(8):1541-1550. doi: 10.1016/j.cgh.2018.11.035. Epub 2018 Nov 23. PMID 30476584
- [Derived] Winthrop KL, Melmed GY, Vermeire S, Long MD, Chan G, Pedersen RD, Lawendy N, Thorpe AJ, Nduaka CI, Su C. Herpes Zoster Infection in Patients With Ulcerative Colitis Receiving Tofacitinib. Inflamm Bowel Dis. 2018 Sep 15;24(10):2258-2265. doi: 10.1093/ibd/izy131. PMID 29850873
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921139&StudyName=Long-Term%20Study%20Of%20CP-690%2C550%20In%20Subjects%20With%20Ulcerative%20Colitis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled in this Study A3921139: 1) who had completed or had early withdrawal due to treatment failure in Study A3921096 (NCT01458574) 2) or who were non-responders after completing induction studies A3921094 (NCT01465763) or A3921095 (NCT01458951). Eligible participants assigned to either Tofacitinib 5 mg BID or 10 mg BID depending if participant was in remission at baseline of A3921139. Remission=total Mayo score <=2 with no individual sub score >1, rectal bleeding sub score =0.
Pre-assignment Details: Treatment failure for Study A3921096 was an increase in Mayo score of >=3 points from baseline value, with an increase in rectal bleeding sub score by >=1 point, and an increase of endoscopic sub score of >=1 point after a minimum of 8 weeks treatment. If endoscopic sub score and baseline endoscopic sub score was 3 (maximum value), then an increase by >=1 point was not needed for treatment failure. But all other components of the treatment failure criteria were needed to be met.
Groups:
- Tofacitinib 5 mg BID: Participants who completed Study A3921096 and were in remission at Week 52 of Study A3921096, received Tofacitinib 5 milligram (mg) tablets twice daily (BID) for maximum of 80 months in this Study A3921139.
- Tofacitinib 10 mg BID: Participants who had completed Study A3921096 and not in remission, or who had early withdrawal due to treatment failure from Study A3921096, or who were non responders after completing A3921094 or A3921095 received Tofacitinib 10 mg tablets twice daily for maximum of 84 months in this Study A3921139.
Period: Overall Study
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Started | 175 | 769
Completed | 91 | 104
Not Completed | 84 | 665
Not completed — Adverse Event | 20 | 80
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 20 | 326
Not completed — Lost to Follow-up | 2 | 5
Not completed — Did not meet entrance criteria | 0 | 1
Not completed — Pregnancy | 2 | 10
Not completed — Protocol Violation | 2 | 7
Not completed — Withdrawal by Subject | 24 | 79
Not completed — Other | 14 | 156

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study medication in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Total
Number analyzed (Participants) | 175 | 769 | 944
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (14.6) | 40.5 (13.5) | 41.2 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 310 | 389
  Male | 96 | 459 | 555
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 136 | 615 | 751
  Black | 0 | 9 | 9
  Asian | 25 | 97 | 122
  Other | 9 | 24 | 33
  Unspecified | 5 | 24 | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 81 months for Tofacitinib 5 mg BID group and up to 85 months for Tofacitinib 10 mg BID group that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and all non-serious AEs.
Time Frame: Baseline up to 28 days after last dose of study drug (up to 81 months for Tofacitinib 5 mg BID group and up to 85 months for Tofacitinib 10 mg BID group)
Population: Safety analysis set (SAS) included all participants who received at least 1 dose of study medication in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 769
Participants
  Participants with AEs | 154 | 626
  Participants with SAEs | 39 | 147

2. Primary Outcome: Number of Participants With Serious Infections as Treatment Emergent Adverse Events (TEAEs)
Description: Serious infections were treated infections that required parenteral antimicrobial therapy or hospitalization for treatment or; met other criteria that required the infection to be classified as a serious adverse event (SAE). SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 81 months for Tofacitinib 5 mg BID group and up to 85 months for Tofacitinib 10 mg BID group that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: as for outcome 1
Population: SAS included all participants who received at least 1 dose of study medication in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 769
Participants | 8 | 31

3. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory abnormalities: Hemoglobin, hematocrit, RBC: <0.8* LLN; reticulocytes (absolute [Abs], %): <0.5* LLN, >1.5* ULN; MCV, MCH: <0.9* LLN, >1.1* ULN; platelets:<0.5* LLN, >1.75* ULN; WBC:<0.6* LLN,>1.5* ULN; lymphocytes (Abs, %), total neutrophils (Abs,%):<0.8* LLN, >1.2* ULN; Basophils (Abs,%),eosinophils(Abs, %),monocytes(Abs, %):>1.2* ULN; total bilirubin,direct bilirubin,indirect bilirubin:>1.5* ULN; AST,ALT,gamma GT, LDH,ALP: >3.0* ULN; total protein,albumin: <0.8* LLN,>1.2* ULN: BUN,creatinine: >1.3* ULN;uric acid:>1.2* ULN; cholesterol,triglycerides: >1.3* ULN; cholesterol (HDL: <0.8* LLN; LDL: >1.2* ULN); sodium: <0.95* LLN, >1.05* ULN; potassium, chloride, calcium, bicarbonate: <0.9* LLN, >1.1* ULN; glucose: <0.6* LLN; creatine kinase >2.0* ULN; urine specific gravity: <1.003; urine pH: <4.5; urine (glucose,protein,blood,nitrite,leukocyte,esterase): >=1; Urine (RBC,WBC): >=20; urine epithelial cells:>=6; urine (casts,granular casts,hyaline casts): >1; urine bacteria:>20.
Time Frame: as for outcome 1
Population: SAS included all participants who received at least 1 dose of study medication in this study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 761
Participants | 162 | 670

4. Primary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Vital sign abnormalities included greater than or equal to (>=) 30 millimeter of mercury [mmHg] increase in systolic blood pressure (BP), >=30 mmHg decrease in systolic BP, Systolic BP (less than [<] 90 mmHg), >=20 mmHg increase in diastolic BP, >=20 mmHg decrease in diastolic BP, diastolic BP (<50 mmHg), pulse rate (<40 beats per minute [BPM]), pulse rate (greater than [>] 120 BPM).
Time Frame: as for outcome 1
Population: SAS included all participants who received at least 1 dose of study medication in this study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable at each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 763
Participants
  Systolic BP (>=30 mmHg increase): number analyzed (Participants) | 172 | 748
  Systolic BP (>=30 mmHg increase) | 20 | 113
  Systolic BP (>=30 mmHg decrease): number analyzed (Participants) | 172 | 748
  Systolic BP (>=30 mmHg decrease) | 19 | 44
  Systolic BP (<90 mmHg) | 3 | 13
  Diastolic BP (>=20 mmHg increase): number analyzed (Participants) | 172 | 748
  Diastolic BP (>=20 mmHg increase) | 21 | 137
  Diastolic BP (>=20 mmHg decrease): number analyzed (Participants) | 172 | 748
  Diastolic BP (>=20 mmHg decrease) | 37 | 78
  Diastolic BP (<50 mmHg) | 3 | 16
  Pulse Rate (<40 BPM) | 1 | 0
  Pulse Rate (>120 BPM) | 0 | 8

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examinations From Baseline
Description: Physical examinations included weight, general appearance, head, ears, eyes, nose, mouth, throat, thyroid, skin (presence of rash), lungs (auscultation), heart (auscultation for presence of murmurs, gallops, rubs, peripheral edema), abdominal (palpation and auscultation), perianal, musculoskeletal, extremities, neurologic (mental status, gait, reflexes, motor and sensory function, coordination) and lymph nodes. Clinically significant changes were judged by the investigator.
Time Frame: as for outcome 1
Population: SAS included all participants who received at least 1 dose of study medication in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 769
Participants | 84 | 391

6. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG abnormalities criteria: maximum PR interval (>=300 millisecond); maximum QRS complex (>=200 millisecond); and maximum QT interval (>=500 millisecond).
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 158 | 707
Participants
  Maximum PR interval (>=300): number analyzed (Participants) | 157 | 706
  Maximum PR interval (>=300) | 0 | 0
  Maximum QRS complex (>=200) | 0 | 0
  Maximum QT interval (>=500) | 0 | 0

7. Primary Outcome: Incidence Rates for Adjudicated Cardiovascular, Malignancy, Opportunistic Infections and Thromboembolic Safety Events
Description: Incidence rates for adjudicated cardiovascular (major adverse cardiovascular event [MACE]), malignancy (non-melanoma skin cancer [NMSC], malignancies excluding NMSC, opportunistic infections (OIs) (both herpes zoster and non herpes zoster OIs) and thromboembolic (venous thromboembolism) safety events were analyzed. This outcome measure was measured in participants with events per 100 participants-years (pt with events/100 pts-yrs).
Time Frame: as for outcome 1
Population: SAS included all participants who received at least 1 dose of study medication in this study.
Measure: Number (95% Confidence Interval); unit: pt with events/100 pts-yrs
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 769
pt with events/100 pts-yrs
  Major adverse cardiovascular event (MACE) | 0.31 [0.04 to 1.13] | 0.11 [0.01 to 0.40]
  Nonmelanoma skin cancer (NMSC) | 0.96 [0.35 to 2.08] | 0.68 [0.35 to 1.19]
  Malignancies excluding NMSC | 1.09 [0.44 to 2.25] | 1.00 [0.60 to 1.59]
  Herpes Zoster OI | 0.47 [0.10 to 1.37] | 0.79 [0.43 to 1.32]
  Non Herpes Zoster OIs | 0.16 [0.00 to 0.87] | 0.17 [0.03 to 0.49]
  Venous thromboembolism | 0.00 [0.00 to 0.57] | 0.33 [0.12 to 0.73]

8. Secondary Outcome: Number of Participants in Remission at Months 2, 12, 24 and 36: Observed Cases
Description: Remission in participants was defined as a total Mayo score of less than or equals to (<=) 2, with no individual sub score exceeding 1 point and a rectal bleeding sub score of 0. Mayo score was an instrument designed to measure disease activity of ulcerative colitis (UC). It consisted of 4 sub scores: stool frequency, rectal bleeding, findings of flexible sigmoidoscopy and physician global assessment (PGA), each sub score graded from 0 to 3 with higher scores indicated higher disease severity. These sub scores were summed up to give a total Mayo score range of 0 to 12, where higher score indicated more severe disease.
Time Frame: Months 2, 12, 24 and 36
Population: FAS included all participants who received at least 1 dose of study medication in this study. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number analyzed" signifies participants evaluable at each specified time point. Data is presented for observed cases, no imputation technique was applied.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 164 | 676
Participants
  Month 2 | 131 | 188
  Month 12: number analyzed (Participants) | 154 | 447
  Month 12 | 129 | 279
  Month 24: number analyzed (Participants) | 132 | 371
  Month 24 | 103 | 264
  Month 36: number analyzed (Participants) | 113 | 299
  Month 36 | 98 | 239

9. Secondary Outcome: Number of Participants in Remission at Months 2, 12, 24 and 36: Non-responder Imputation- Last Observation Carried Forward (NRI-LOCF)
Description: Remission in participants was defined as a total Mayo score of <=2, with no individual sub score exceeding 1 point and a rectal bleeding sub score of 0. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 sub scores: stool frequency, rectal bleeding, findings of flexible sigmoidoscopy and PGA, each sub score graded from 0 to 3 with higher scores indicated higher disease severity. These sub scores were summed up to give a total Mayo score range of 0 to 12, where higher score indicated more severe disease.
Time Frame: Months 2, 12, 24 and 36
Population: FAS included all participants who received at least 1 dose of study medication in this study. NRI method was used for missing data except for visits after a participant advanced to other studies where LOCF method was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 769
Participants
  Month 2 | 131 | 188
  Month 12 | 129 | 279
  Month 24 | 103 | 264
  Month 36 | 103 | 259

10. Secondary Outcome: Number of Participants in Clinical Remission at Months 2, 12, 24 and 36: Observed Cases
Description: Clinical remission in participants was defined as a total Mayo score of <=2 with no individual sub score exceeding 1 point. Mayo score was an instrument designed to measure disease activity of UC. It consisted of 4 sub scores: stool frequency, rectal bleeding, findings of flexible sigmoidoscopy and PGA, each graded from 0 to 3 with higher scores indicated higher disease severity. These sub scores were summed up to give a total Mayo score range of 0 to 12, where higher score indicated more severe disease.
Time Frame: Months 2, 12, 24 and 36
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 164 | 676
Participants
  Month 2 | 132 | 191
  Month 12: number analyzed (Participants) | 154 | 447
  Month 12 | 129 | 282
  Month 24: number analyzed (Participants) | 132 | 371
  Month 24 | 104 | 266
  Month 36: number analyzed (Participants) | 113 | 299
  Month 36 | 102 | 240

11. Secondary Outcome: Number of Participants in Clinical Remission at Months 2, 12, 24 and 36: Non-responder Imputation- Last Observation Carried Forward (NRI-LOCF)
Description: as for outcome 10
Time Frame: Months 2, 12, 24 and 36
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 769
Participants
  Month 2 | 132 | 191
  Month 12 | 129 | 282
  Month 24 | 104 | 266
  Month 36 | 107 | 260

12. Secondary Outcome: Number of Participants in Partial Mayo Score (PMS) Remission at Months 1, 4, 6, 9, 15, 18, 21, 27, 30, 33, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69, 72, 75, 78, 81 and 84: Observed Cases
Description: PMS was an instrument designed to measure disease activity of UC without endoscopy. It consisted of 3 sub scores: stool frequency, rectal bleeding and PGA, each sub score graded from 0 to 3 with higher scores indicated higher disease severity. These sub scores were summed up to give a total score range of 0 to 9, where higher score indicated more severe disease. PMS remission was defined as a partial Mayo score <=2 with no individual sub score >1.
Time Frame: Months 1, 4, 6, 9, 15, 18, 21, 27, 30, 33, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69, 72, 75, 78, 81 and 84
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 166 | 729
Participants
  Month 1 | 158 | 275
  Month 4: number analyzed (Participants) | 165 | 532
  Month 4 | 152 | 375
  Month 6: number analyzed (Participants) | 166 | 505
  Month 6 | 155 | 395
  Month 9: number analyzed (Participants) | 160 | 469
  Month 9 | 154 | 390
  Month 15: number analyzed (Participants) | 145 | 418
  Month 15 | 139 | 361
  Month 18: number analyzed (Participants) | 144 | 404
  Month 18 | 137 | 354
  Month 21: number analyzed (Participants) | 138 | 394
  Month 21 | 125 | 351
  Month 27: number analyzed (Participants) | 125 | 348
  Month 27 | 117 | 319
  Month 30: number analyzed (Participants) | 124 | 338
  Month 30 | 117 | 307
  Month 33: number analyzed (Participants) | 118 | 326
  Month 33 | 111 | 304
  Month 39: number analyzed (Participants) | 105 | 281
  Month 39 | 102 | 261
  Month 42: number analyzed (Participants) | 100 | 253
  Month 42 | 95 | 236
  Month 45: number analyzed (Participants) | 102 | 226
  Month 45 | 95 | 212
  Month 48: number analyzed (Participants) | 92 | 199
  Month 48 | 87 | 183
  Month 51: number analyzed (Participants) | 89 | 175
  Month 51 | 87 | 162
  Month 54: number analyzed (Participants) | 71 | 147
  Month 54 | 68 | 140
  Month 57: number analyzed (Participants) | 56 | 128
  Month 57 | 54 | 120
  Month 60: number analyzed (Participants) | 39 | 107
  Month 60 | 38 | 98
  Month 63: number analyzed (Participants) | 28 | 89
  Month 63 | 28 | 80
  Month 66: number analyzed (Participants) | 21 | 73
  Month 66 | 19 | 67
  Month 69: number analyzed (Participants) | 11 | 54
  Month 69 | 10 | 49
  Month 72: number analyzed (Participants) | 6 | 44
  Month 72 | 6 | 40
  Month 75: number analyzed (Participants) | 3 | 26
  Month 75 | 3 | 24
  Month 78: number analyzed (Participants) | 4 | 19
  Month 78 | 4 | 18
  Month 81: number analyzed (Participants) | 0 | 11
  Month 81 |  | 10
  Month 84: number analyzed (Participants) | 0 | 8
  Month 84 |  | 6

13. Secondary Outcome: Number of Participants in Partial Mayo Score (PMS) Remission at Months 1, 4, 6, 9, 15, 18, 21, 27, 30, 33, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69, 72, 75, 78, 81 and 84: Non-responder Imputation- Last Observation Carried Forward (NRI-LOCF)
Description: PMS was an instrument designed to measure disease activity of UC without endoscopy. It consisted of 3 sub scores: stool frequency, rectal bleeding and PGA, each sub score graded from 0 to 3 with higher scores indicated higher disease severity. These sub scores were summed up to give a total PMS score range of 0 to 9, where higher score indicated more severe disease. PMS remission was defined as a partial Mayo score <=2 with no individual sub score >1.
Time Frame: Months 1, 4, 6, 9, 15, 18, 21, 27, 30, 33, 39, 42, 45, 48, 51, 54, 57, 60, 63, 66, 69, 72, 75, 78, 81 and 84
Population: FAS included all participants who received at least 1 dose of study medication in this study. Here, "Number analyzed" signifies participants evaluable at each specified time point. NRI method was used for missing data at all visits except for visits after a participant advanced to other studies and would reach the visits if the participant stayed in the study where LOCF method was used.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 769
Participants
  Month 1 | 158 | 275
  Month 4 | 152 | 375
  Month 6 | 155 | 395
  Month 9 | 154 | 390
  Month 15 | 139 | 361
  Month 18 | 137 | 354
  Month 21 | 125 | 351
  Month 27 | 117 | 325
  Month 30 | 117 | 316
  Month 33 | 114 | 317
  Month 39 | 108 | 293
  Month 42 | 102 | 286
  Month 45 | 102 | 283
  Month 48 | 95 | 274
  Month 51 | 96 | 267
  Month 54: number analyzed (Participants) | 170 | 764
  Month 54 | 76 | 250
  Month 57: number analyzed (Participants) | 160 | 753
  Month 57 | 61 | 234
  Month 60: number analyzed (Participants) | 149 | 732
  Month 60 | 44 | 213
  Month 63: number analyzed (Participants) | 135 | 707
  Month 63 | 31 | 194
  Month 66: number analyzed (Participants) | 125 | 659
  Month 66 | 22 | 168
  Month 69: number analyzed (Participants) | 114 | 562
  Month 69 | 13 | 131
  Month 72: number analyzed (Participants) | 109 | 468
  Month 72 | 7 | 102
  Month 75: number analyzed (Participants) | 102 | 412
  Month 75 | 3 | 73
  Month 78: number analyzed (Participants) | 96 | 339
  Month 78 | 4 | 52
  Month 81: number analyzed (Participants) | 95 | 284
  Month 81 | 0 | 29
  Month 84: number analyzed (Participants) | 91 | 210
  Month 84 | 0 | 15

14. Secondary Outcome: Number of Participants Who Achieved Mucosal Healing at Months 2, 12, 24 and 36: Observed Cases
Description: Mucosal healing in participants was defined as Mayo endoscopic sub score of 0 or 1. The Mayo endoscopic sub score consisted of the findings of flexible sigmoidoscopy, graded from 0 to 3 with higher sub scores indicated higher disease severity.
Time Frame: Months 2, 12, 24 and 36
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 169 | 690
Participants
  Month 2 | 152 | 279
  Month 12: number analyzed (Participants) | 156 | 458
  Month 12 | 140 | 340
  Month 24: number analyzed (Participants) | 136 | 382
  Month 24 | 119 | 307
  Month 36: number analyzed (Participants) | 115 | 307
  Month 36 | 107 | 265

15. Secondary Outcome: Number of Participants Who Achieved Mucosal Healing at Months 2, 12, 24 and 36: Non-responder Imputation- Last Observation Carried Forward (NRI-LOCF)
Description: Mucosal healing in participants was defined as mayo endoscopic sub score of 0 or 1. The mayo endoscopic sub score consisted of the findings of flexible sigmoidoscopy, graded from 0 to 3 with higher sub scores indicating higher disease severity.
Time Frame: Months 2, 12, 24 and 36
Population: FAS included all participants who received at least 1 dose of study medication in this study. NRI method was used for missing data at all visits and LOCF method was used for visits after a participant advanced to next study.
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 769
Participants
  Month 2 | 152 | 279
  Month 12 | 140 | 340
  Month 24 | 119 | 307
  Month 36 | 113 | 285

16. Secondary Outcome: Number of Participants With Total Inflammatory Bowel Disease Questionnaire (IBDQ) Score >=170 at Months 2, 6, 12, 18, 24, 30, 36, 48, 60, 72 and 84: Non-responder Imputation- Last Observation Carried Forward (NRI-LOCF)
Description: IBDQ was a psychometrically validated patient reported outcome (PRO) instrument for measuring the disease-specific quality of life in participants with inflammatory bowel disease (IBD), including ulcerative colitis consisted of 32 items scored from 1 (worst response) to 7 (best response). For each domain, higher score indicates better quality of life (QOL). Total IBDQ score was the sum of each item score, and ranged from 32 to 224 with a higher score indicated better QOL.
Time Frame: Months 2, 6, 12, 18, 24, 30, 36, 48, 60, 72 and 84
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 175 | 769
Participants
  Month 2 | 154 | 419
  Month 6 | 151 | 395
  Month 12 | 140 | 365
  Month 18 | 123 | 354
  Month 24 | 120 | 315
  Month 30 | 115 | 299
  Month 36 | 111 | 294
  Month 48 | 93 | 265
  Month 60: number analyzed (Participants) | 149 | 732
  Month 60 | 45 | 215
  Month 72: number analyzed (Participants) | 109 | 468
  Month 72 | 8 | 99
  Month 84: number analyzed (Participants) | 91 | 210
  Month 84 | 0 | 14

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose of study drug (up to 81 months for Tofacitinib 5 mg BID group and up to 85 months for Tofacitinib 10 mg BID group)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Analysis performed on safety analysis set.
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
All-Cause Mortality (participants affected / at risk) | 0/175 | 6/769
Serious Adverse Events (participants affected / at risk) | 39/175 | 147/769
Other Adverse Events (participants affected / at risk) | 134/175 | 550/769
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5 mg BID (N=175) | Tofacitinib 10 mg BID (N=769)
Anaemia (Blood and lymphatic system disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Thyroid mass (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal skin tags (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 4 | 38
Colon dysplasia (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Megacolon (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 0 | 3
Arthritis bacterial (Infections and infestations) | 0 | 1
Atypical pneumonia (Infections and infestations) | 0 | 1
Bacterial vaginosis (Infections and infestations) | 1 | 0
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Complicated appendicitis (Infections and infestations) | 1 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 4
Herpes zoster meningitis (Infections and infestations) | 0 | 1
Histoplasmosis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Meningitis viral (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 2
Osteomyelitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 0 | 1
Pulmonary mycosis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epstein-Barr virus associated lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 0 | 1
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Device loosening (Product Issues) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 2
Prerenal failure (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 2
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Eosinophilic pustular folliculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib 5 mg BID (N=175) | Tofacitinib 10 mg BID (N=769)
Anaemia (Blood and lymphatic system disorders) | 3 | 36
Lymphopenia (Blood and lymphatic system disorders) | 6 | 13
Abdominal pain (Gastrointestinal disorders) | 6 | 47
Abdominal pain upper (Gastrointestinal disorders) | 4 | 24
Colitis ulcerative (Gastrointestinal disorders) | 44 | 131
Constipation (Gastrointestinal disorders) | 7 | 20
Diarrhoea (Gastrointestinal disorders) | 9 | 34
Dyspepsia (Gastrointestinal disorders) | 8 | 12
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 15
Haemorrhoids (Gastrointestinal disorders) | 3 | 20
Nausea (Gastrointestinal disorders) | 1 | 30
Vomiting (Gastrointestinal disorders) | 3 | 20
Fatigue (General disorders) | 5 | 33
Oedema peripheral (General disorders) | 4 | 13
Pyrexia (General disorders) | 2 | 25
Bronchitis (Infections and infestations) | 17 | 30
Ear infection (Infections and infestations) | 4 | 6
Gastroenteritis (Infections and infestations) | 12 | 51
Herpes zoster (Infections and infestations) | 12 | 50
Influenza (Infections and infestations) | 23 | 63
Latent tuberculosis (Infections and infestations) | 4 | 13
Nasopharyngitis (Infections and infestations) | 41 | 157
Oral herpes (Infections and infestations) | 1 | 18
Pharyngitis (Infections and infestations) | 8 | 14
Pneumonia (Infections and infestations) | 4 | 9
Rhinitis (Infections and infestations) | 5 | 7
Sinusitis (Infections and infestations) | 8 | 25
Upper respiratory tract infection (Infections and infestations) | 19 | 77
Urinary tract infection (Infections and infestations) | 13 | 34
Viral upper respiratory tract infection (Infections and infestations) | 5 | 7
Ligament sprain (Injury, poisoning and procedural complications) | 4 | 8
Skin laceration (Injury, poisoning and procedural complications) | 5 | 4
Alanine aminotransferase increased (Investigations) | 6 | 11
Aspartate aminotransferase increased (Investigations) | 5 | 8
Blood cholesterol increased (Investigations) | 7 | 18
Blood creatine phosphokinase increased (Investigations) | 19 | 85
Lymphocyte count decreased (Investigations) | 3 | 18
White blood cell count decreased (Investigations) | 4 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 38
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 76
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 28
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 10
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 9
Tendonitis (Musculoskeletal and connective tissue disorders) | 5 | 4
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 14
Dizziness (Nervous system disorders) | 4 | 14
Headache (Nervous system disorders) | 12 | 57
Paraesthesia (Nervous system disorders) | 2 | 17
Anxiety (Psychiatric disorders) | 6 | 16
Depression (Psychiatric disorders) | 4 | 12
Insomnia (Psychiatric disorders) | 5 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 38
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Acne (Skin and subcutaneous tissue disorders) | 5 | 20
Rash (Skin and subcutaneous tissue disorders) | 4 | 38
Hypertension (Vascular disorders) | 17 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/12/NCT01470612/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT01470612/SAP_001.pdf